CLINICAL TRIAL: NCT05925491
Title: Neoadjuvant Pembrolizumab Plus Chemotherapy in Locally Advanced Sinonasal Carcinoma
Brief Title: Pembrolizumab in Locally Advanced Sinonasal Carcinoma
Acronym: NeoPeSino
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoPeSino
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Sinonasal Undifferentiated Carcinoma
Keywords: Sinonasal Undifferentiated Carcinoma; SNUC; neoadjuvant immunotherapy; neoadjuvant treatment; locally advanced; pembrolizumab; neoadjuvant
MeSH Terms: conditions — Sinonasal undifferentiated carcinoma | interventions — pembrolizumab; Cisplatin; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant Pembrolizumab (Experimental): Patients will receive pembrolizumab 200 mg + cisplatin 75mg/mq (or Carboplatin AUC 5) and docetaxel 75 mg/mq every three weeks (Q3W) for 3 courses, followed by standard of care.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administration in combination with chemotherapy for 3 cycles, followed by standard of care
Drug: Cisplatin — Cisplatin 75mg/mq in combination with pembrolizumab 200 mg and docetaxel 75 mg/mq every three weeks (Q3W) for 3 courses.
Drug: Docetaxel — Docetaxel 75 mg/mq in combination with pembrolizumab 200 mg and cisplatin 75 mg/mq every three weeks (Q3W) for 3 courses.
Drug: Carboplatin — Carboplatin AUC 5 alternative to Cisplatin if toxicities occur.

SUMMARY:
This study will test the Safety and activity of pembrolizumab plus chemotherapy as neoadjuvant treatment in locally advanced sinonasal undifferentiated carcinoma (SNUC).

Activity of neoadjuvant chemotherapy in locally advanced SNUC has been already demonstrated; the primary hypothesis is that the addition of pembrolizumab as neoadjuvant and adjuvant agent might confirm the results obtained with a combined treatment strategy including chemotherapy, decreasing the burden of treatment-related side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Have centrally histologically-confirmed, treatment-naïve SNUC that is considered curable by local therapies.
2. Have locally advanced disease defined as stage III of IV a-b according to American Joint Committee on Cancer (AJCC) cancer staging system VIII edition.
3. Be willing and able to provide written informed consent for the trial. The subject may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
4. Be ≥ 18 years of age on day of signing informed consent.
5. Have measurable disease based on RECIST 1.1 as determined by the site.
6. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
7. Demonstrate adequate organ function.
8. A male participant must agree to use contraception during the treatment period and for at least 180 days after last dose, corresponding to time needed to eliminate any study treatments plus an additional 90 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity. He must refrain from donating sperm during this period, too.
9. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   o Not a woman of childbearing potential (WOCBP) OR a WOCBP who agrees use contraception during the treatment period and for at least 180 days (corresponding to time needed to eliminate any study treatments plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment.
10. Have provided tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has disease that is deemed not suitable for local therapy administered with curative intent (e.g. severe brain involvement).
2. 2. Have metastatic disease defined as stage IV c according to AJCC cancer staging system VIII edition.
3. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
5. Has received prior systemic anti-cancer therapy including investigational agents prior to allocation.
6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. Administration of killed vaccines is allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ (eg, breast carcinoma or cervical cancer in situ that have undergone potentially curative therapy are not excluded
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
11. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
13. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
14. Has an active infection requiring systemic therapy.
15. Has a known history of Human Immunodeficiency Virus (HIV) infection.
16. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA qualitative is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
17. Has a known history of active TB (Bacillus Tuberculosis).
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Neoadjuvant therapy objective response rate (ORR) | Up to 24 months after the end of neoadjuvant treatment
  ORR defined as the sum of complete remission (CRs) and partial responses (PRs) by RECIST v. 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Locati, MD, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No